CLINICAL TRIAL: NCT00133068
Title: Collaboration to Reduce Disparities in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government); Dickinson College (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Stephen E. Kimmel, Stephen E. Kimmel, M.D., M.S.C.E,, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 707850
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Health Behaviors; Patient Compliance
MeSH Terms: conditions — Hypertension; Health Behavior; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Control
  Interventions: Behavioral: Control
- 2 (Experimental): Reduction of financial barrier
  Interventions: Behavioral: Reduction in financial barrier
- 3 (Experimental): Computer Intervention
  Interventions: Behavioral: Computer
- 4 (Experimental): Reduction of financial barrier and Computer Intervention
  Interventions: Behavioral: Computer intervention & reduction of financial barrier

INTERVENTIONS:
Behavioral: Computer — Computer intervention only
  Arms: 3
Behavioral: Reduction in financial barrier — Copay only
  Arms: 2
Behavioral: Computer intervention & reduction of financial barrier — computer intervention & copay
  Arms: 4
Behavioral: Control — No intervention
  Arms: 1

SUMMARY:
A large number of African-American and low socioeconomic patients have poorly controlled high blood pressure because of not being able to take their high blood pressure medications. This puts these patients at higher risk of heart and kidney disease, stroke and death. This study is designed to reduce the barriers that prevent patients from taking their high blood pressure medications.

DETAILED DESCRIPTION:
The objective of this study is to determine the effectiveness and cost-effectiveness of two interventions aimed at reducing barriers to blood pressure (BP) control in an indigent and African-American population. Specifically, we will conduct a randomized controlled trial comparing BP control using either: (1) reimbursing patients for filling prescriptions (reimbursement arm); (2) a computer-based behavioral intervention (behavioral arm); (3) both the reimbursement and behavioral arms (combined arms); or (4) neither.

The ultimate goal of this study is to reduce the incidence of HTN-related CVD among these populations thereby reducing cardiovascular health disparities. Specific aims of the study are to:

1. test whether receiving money each time the patient fills a prescription for medications improves BP control by a clinically significant amount.

   H1: Reimbursing patients for filling prescriptions will significantly improve BP control.
2. test whether a computer-based behavioral intervention improves BP control by a clinically significant amount.

   H2: A computer-based behavioral intervention will significantly improve BP control.
3. test whether the two interventions are more effective in improving BP control than either alone.

   H3: The effect of improving BP control of administering both interventions together will be greater than the sum of the individual effects of each intervention alone.
4. examine the relative cost effectiveness of reimbursement for filling prescriptions, a computer-based behavioral intervention, and the combination of the two.

H4: Both interventions will be cost-effective relative to other commonly-covered services.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Philadelphia Veterans Administration Hospital Primary Care Clinic, PinnacleHealth Adult Outpatient Clinics and the VA Pittsburgh Healthcare System who have a diagnosis of hypertension; are currently taking antihypertensive medications; and have elevated blood pressure.

Exclusion Criteria:

* Under 21 years of age
* Have a diagnosis of:

  * Atrial fibrillation;
  * Metastatic cancer;
  * End stage renal disease (ESRD) with dialysis;
  * Dementia;
  * New York Heart Association (NYHA) class IV congestive heart failure (CHF);
  * Blind or deaf;
  * Other reason for life expectancy of less than 1 year.
* Are currently participating in another experimental study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 months

SECONDARY OUTCOMES:
Cost | 12 months
Blood pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Kimmel, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - PinnacleHealth Adult Outpatient Clinics, Harrisburg, Pennsylvania
  - Veterans Administration Medical Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Volpp KG, Troxel AB, Long JA, Ibrahim SA, Appleby D, Smith JO, Jaskowiak J, Helweg-Larsen M, Doshi JA, Kimmel SE. A randomized controlled trial of co-payment elimination: the CHORD trial. Am J Manag Care. 2015 Aug;21(8):e455-64. PMID 26625505